CLINICAL TRIAL: NCT05100420
Title: Hearts in Rhythm Organization Hypertrophic Cardiomyopathy Registry, Biobank and Imaging Data Repository (HiRO-HCM)
Brief Title: Hypertrophic Cardiomyopathy Registry, Biobank and Imaging Data Repository
Acronym: HiRO-HCM
Status: Enrolling by invitation | Type: Observational
Sponsor: Montreal Heart Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Rafik Tadros, Cardiologist, Clinician Scientist, Montreal Heart Institute
Other Study IDs: MP-33-2021-2872
Record Dates: First submitted 2021-10-18; First posted 2021-10-29 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Hypertrophic Cardiomyopathy; Hypertrophic Obstructive Cardiomyopathy; Familial Hypertrophic Cardiomyopathy; Cardiomyopathies
Keywords: Genetics; Echocardiography; Cardiac magnetic resonance imaging; Biomarker; Sudden cardiac death; Genome-wide association study; Risk prediction model
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Cardiomyopathy, Hypertrophic, Familial; Cardiomyopathies; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — DNA isolated from blood or saliva Plasma Myocardial tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Hearts in Rhythm Organization (HiRO) is a national network of Canadian researchers/clinicians, working towards a better understanding of the rare genetic causes of sudden cardiac death (SCD). The HiRO Hypertrophic Cardiomyopathy registry, biobank and imaging data repository (HiRO-HCM) is a multicenter study that will prospectively enroll patients with HCM as well as those carrying sarcomeric gene variants predisposing to HCM.

The objectives of HiRO-HCM are:

1. to better understand the natural history of the disease and identify clinical markers and biomarkers for adverse outcomes;
2. to derive and validate risk prediction models for disease expression, complications and response to therapy;
3. to better define the genetic architecture of sarcomeric and non-sarcomeric HCM.

DETAILED DESCRIPTION:
PATIENT ENROLLMENT:

Eligible patients will be included from HiRO sites or collaborating centres. Patients will be contacted by the local investigator or a research coordinator. Willing individuals will be interviewed by the research coordinator and given information about HiRO-HCM. The consent form will be reviewed and discussed with the coordinator. The investigators will also be available for any questions that the coordinator is unable to answer. Potential participants will have sufficient time to consider participating in HiRO-HCM. Written informed consent will be obtained from eligible patients or legal guardians. Participants will be able to withdraw their participation at any time.

BASELINE DATA COLLECTION:

Clinical data will be collected from willing/consented registry participants. All demographic and medical information pertaining to the cardiac history and comorbidities of eligible patients will be collected at baseline, including clinical information, diagnostic test results, genetic testing results, family history and ethnicity, as well as current and previous treatments. Healthcare information will be coded in compliance with Canada's Tri-Council Policy Statement criteria: direct identifiers will be removed and replaced with a unique study code that does not use personal information such as the participant's health number, social insurance number or name. The coded data will be transferred into the clinical research database using a web-based electronic case report form (eCRF), using REDcap. The clinical research database will be managed by the Montreal Health Innovations Coordinating Center (MHICC; mhicc.org). Study participants will be identified by subject number only (research HiRO-HCM ID). The research ID uniquely identifying each subject eCRF within the database will be attributed in REDcap but the master list of registry participants with their study identifiers will be kept separately from the clinical research database. This master list will be stored in an encrypted file within the research office of each site investigators under their supervision. Only the site investigators and their local research staff will have access to this list.

BIOSPECIMEN COLLECTION:

Consented participants will undergo biosampling at enrollment for the primary purpose of DNA isolation and genetic studies. The preferred biosampling method is blood sampling using a standard venipuncture. Blood sampling allows for high quality DNA extraction as well as collection of plasma for future circulating biomarkers studies. As an alternative to blood sampling, collection of saliva using DNA genotek kits, or equivalent, is allowed in the following contexts:

* Patient enrollment is performed remotely. This is particularly relevant in the context of the ongoing SARS-CoV-2 pandemic, where physical distancing is preferred.
* Patient is a child <14 years old without planned clinically indicated blood sampling.

Participants for which saliva collection is chosen should be made aware of the possibility to request a blood sample in the future.

The HiRO-HCM biobank will be directed by the Beaulieu-Saucier Pharmacogenomics Center (PGx; http://www.pharmacogenomics.ca), operating under Good Laboratory/Clinical Practices (GLP/GCP) standards.

DNA isolation and long-term storage will be done at PGx, while long-term storage of plasma samples will be done at the MHI research center, in dedicated freezers located in a room with restricted access. Samples of subjects that withdraw their participation will be destroyed.

IMAGING DATA TRANSFER:

For all consented participants, de-identified transthoracic echocardiography (TTE) and cardiac magnetic resonance (CMR) imaging data will be transferred to the Montreal Heart Institute imaging core-lab for central interpretation and long term storage. At minimum, the following imaging studies are requested:

1. First available TTE
2. First available CMR, preferably with gadolinium injection
3. Last available TTE
4. Last available CMR, preferably with gadolinium injection

For patients that underwent alcohol septal ablation, surgical myectomy and/or cardiac transplantation, the last available TTE and CMR studies prior to all these interventions should also be transferred.

Digital Imaging and Communications in Medicine (DICOM) imaging data will be de-identified prior to transfer. De-identification will be performed at each site, by removing the patient's name and replacing the clinical identification number with the research HiRO-HCM ID. DICOM data will be stored using the Canadian Imaging network infrastructure (canadianimagingnetwork.org).

PATIENT FOLLOW-UP:

Participants with a clinical diagnosis of HCM are expected to undergo yearly clinic visits, as per standard care. Participants without yearly clinic visits will be contacted by phone. Follow-up visits will assess for living status, functional class, as well as for arrhythmic, heart failure and thromboembolic events. Follow-up data will be entered by the local investigator and/or research coordinator into an eCRF managed by the MHICC. De-identified documentation of clinical events including ECG, intracardiac tracing, clinical notes, imaging reports, and procedural reports will be uploaded to the database for centralized ad-hoc event adjudication.

De-identified DICOM images of TTE and CMR studies performed clinically during follow-up will be uploaded to the MHI imaging core-lab similarly as for baseline imaging studies.

For participants that will undergo septal myectomy for drug-refractory obstructive HCM, or cardiac transplantation, surgical tissue samples will be collected using the Qiagen PAXgene tissue preservation system or equivalent, allowing for future somatic DNA, RNA and proteomic analyses. The samples will be stored at the MHI research center.

ELIGIBILITY:
Inclusion Criteria:

Patients with (1) AND/OR (2)

1. Clinical diagnosis of HCM, defined as

   1. maximal LVWT ≥15mm, or
   2. maximal LVWT ≥13mm, in presence of a diagnosis of first degree relative with HCM, or
   3. septal wall thickness with z-score >2 in a child

   AND/OR
2. Carrier of a pathogenic or likely pathogenic genetic variant in a sarcomeric gene (ACTC1, FHOD3, MYBPC3, MYH7, MYL2, MYL3, TNNI3, TNNT2, TPM1). Variant classification should be performed by a certified diagnostic laboratory according to the American College of Medical Genetics and Genomics (ACMG) guidelines.

Exclusion Criteria:

1. Clinical or molecular diagnosis of Noonan syndrome or other Rasopathies
2. Clinical or molecular diagnosis of metabolic disease associated with cardiomyopathy, such as Pompe (GAA), Fabry (GLA), Danon (LAMP2), AMP-kinase (PRKAG2), and carnitine disorders
3. Clinical diagnosis of a neuromuscular disease associated with cardiomyopathy, such as Friedrich's ataxia
4. Clinical diagnosis of cardiac amyloidosis with or without the presence of genetic variants in TTR
5. Clinical or molecular diagnosis of mitochondrial cardiomyopathy
6. Diagnosis of HCM >65 years old AND absence of pathogenic or likely pathogenic variant in a sarcomeric gene (as defined in inclusion criterion 1B above)
7. History of myocardial infarction
8. History of moderate or severe aortic stenosis
9. History of congenital heart defects requiring percutaneous or surgical correction
10. History of severe hypertension defined as a systolic blood pressure >180 mmHg and/or diastolic blood pressure >110 mmHg AND absence of pathogenic or likely pathogenic variant in a sarcomeric gene (as defined in inclusion criterion 1B above)
11. Refusal to provide informed consent or to provide a biospecimen for DNA analysis
12. No possibility to upload transthoracic echocardiogram or cardiac magnetic resonance imaging for core lab interpretation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The HiRO-HCM registry, biobank and imaging data repository is a multicenter collaboration that will prospectively enroll patients with HCM as well as those carrying genetic variants predisposing to HCM.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-02-23 (Actual); Primary Completion 2026-02-23 (Estimated); Study Completion 2027-08-23 (Estimated)

PRIMARY OUTCOMES:
Create a Canadian Research Database, a biobank and an imaging data repository for those affected by hypertrophic cardiomyopathy (HCM) or carrying a sarcomeric gene variant associated with HCM | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Rafik Tadros, Dr., Principal Investigator — Montreal Heart Institute
Locations (13):
- Canada (13):
  - Mazankowski Alberta Heart Institute, Edmonton, Alberta
  - UBC St. Paul's Hospital, Vancouver, British Columbia
  - Vancouver Island Health Authority, Victoria, British Columbia
  - IWK Health Centre, Halifax, Nova Scotia
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - McMaster University, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - Hôpital Ste-Justine, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - Institut Universitaire de Cardiologie et Pneumologie de Québec, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No